CLINICAL TRIAL: NCT04390542
Title: A Pilot Study Evaluating Feasibility, Acceptability, Usability, Satisfaction and Preliminary Efficacy of an Intervention for Caregivers of Patients Undergoing HSCT or CAR T-cell Therapy
Brief Title: Intervention for Caregivers of Patients Undergoing HSCT or CAR T-cell Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE8Z20
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Blood Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation intervention (Experimental): Psychoeducatoinal intervention
  Interventions: Behavioral: Psychoeducation
- Usual care (No Intervention): Information from healthcare providers

INTERVENTIONS:
Behavioral: Psychoeducation — 6 sessions (in-person, videoconference, or phone delivery per the caregiver's choice) between the interventionist and caregivers. Topics covered in sessions include:
  Session 1: Communication, Support, Self Care, Symptom Management
  Sessions 2-4: Communication, Symptom Management, Support
  Sessions 5-6: Self-Care, Symptom Management, Communication, Support, Future Planning
  Arms: Psychoeducation intervention

SUMMARY:
The purpose of this study is to determine which of two approaches is helpful to support caregivers of patients undergoing Hematopoietic Stem Cell Transplant (HSCT) or Chimeric Antigen Receptors (CAR) T-cell therapy at Seidman Cancer Center. This study will take start before you begin treatment until 2 months after your hospital discharge.

DETAILED DESCRIPTION:
This is a two-group, randomized pilot study to test the feasibility, acceptability, usability, satisfaction and preliminary efficacy of a behavioral (psychoeducation) intervention, as compared to a usual care (information from healthcare providers) control group, on caregiver outcomes. The control and intervention groups will receive the standard University Hospitals Seidman Cancer Center (SCC) binder of relevant information regarding care of the patient undergoing HSCT or CAR T-cell therapy. This information will be given to the caregiver by the health care provider. In addition, the intervention group will receive 6 individual sessions with an interventionist during all phases of HSCT or CAR T-cell therapy. The independent variable is group assignment.

The primary objective of this study is to explore the feasibility and acceptability of a psycho-educational intervention designed for caregivers of patients receiving HSCT (allogenic or autologous) or CAR T-cell therapy.

The secondary objective of this study is to explore the usability, satisfaction and preliminary efficacy of a psycho-educational intervention designed for caregivers of patients receiving HSCT (allogenic or autologous) or CAR T-cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Has a diagnosis of blood cancer (leukemia, lymphoma, myeloma, MDS, MPN, CML, CMML) and is scheduled to undergo HCST or CAR T-cell therapy at SCC
  * Will receive HSCT or CAR T-cell therapy and follow-up care from a medical oncologist at University Hospitals Seidman Cancer Center (SCC)
  * Has English as their primary language
  * Provides consent for his/her own treatment and procedures
  * Has an identified caregiver (per SCC-HSCT and CAR T-cell therapy protocol) who will be involved in the patient's care post-HCST or CAR T-cell therapy
* Caregivers

  * An adult family or friend (at least 18 years old) of a patient scheduled to receive HSCT or CAR T-cell therapy at SCC
  * Identifies himself/herself as the caregiver who will be responsible for the patient's care post-HSCT or CAR T-cell therapy
  * Has English as their primary language
  * Is capable of providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Time to identify and recruit dyads in months | 2 months post-hospital discharge, an average of 2 months
  Feasibility, as measured by time to identify and recruit dyads (benchmark 3 months)
Accrual rates | 2 months post-hospital discharge, an average of 2 months
  Feasibility, as measured by accrual rates of eligible participants
Retention rate | 2 months post-hospital discharge, an average of 2 months
  Feasibility, as measured by retention rate
Data collection completion rate | 2 months post-hospital discharge, an average of 2 months
  Feasibility as measured by completion of data collection across study timepoints
Average acceptability scale scores | 2 months post-hospital discharge, an average of 2 months
  Acceptability, as measured by average acceptability scale scores, with overall score ranging from 6-30. According to prior research, a score of 80% of higher (total score of 24 or higher) is considered acceptable for use.
Average System Usability Scale scores | 2 months post-hospital discharge, an average of 2 months
  Usability, as measured by average System Usability Scale scores. This is a 10 item scale scored on a 5 point Likert scale with total summed scores ranging from 0-50. Total scores are multiplied by 2 to produce an overall score ranging from 0-100 with scores > 68 considered to be above average usability.
Mean caregiver satisfaction | 2 months post-hospital discharge, an average of 2 months
  Caregiver satisfaction will be evaluated by having caregivers evaluate their satisfaction with each of the 6 modules at the end of each module. After completing each module, they will be sent via REDCap a single item evaluation scale (0 -10; 0=Not at all satisfied; 10=Highly satisfied). Scores >7 will be considered acceptable. Mean and standard deviation to describe subjects' overall satisfaction with the intervention reported.
End-of-study caregiver satisfaction scores | 2 months post-hospital discharge, an average of 2 months
  End-of-study caregiver satisfaction, as measured by end of study exit interview that assesses overall satisfaction with intervention (Likert Scale). Scores range from 0 to 10, with higher scores indicating more satisfaction.

SECONDARY OUTCOMES:
Caregiver anxiety as measured by PROMISR Short Form v1.0 - Anxiety scores | Baseline, hospital discharge, 2 months post hospital discharge
  Caregiver anxiety as measured by PROMISR Short Form v1.0 - Anxiety scores. Scores range from 1 to 5, with higher scores indicating worse anxiety.
  Evaluated for changes over 3 time points using repeated measures analysis of variance (RMANOVA)-between and within model- controlling for caregiver age, race, and gender
Caregiver Healthcare Related Quality Of Life (HRQOL) | Baseline, hospital discharge, 2 months post hospital discharge
  Caregiver HRQOL, evaluated for changes over 3 time points using repeated measures analysis of variance (RMANOVA)-between and within model- controlling for caregiver age, race, and gender. HRQOL scores range from 1 to 5, with higher scores indicating better outcomes.
Distress as measured by the the NCCN distress thermometer | Baseline, hospital discharge, 2 months post hospital discharge
  Distress as measured by the NCCN distress thermometer. Thermometer scores range from 0 to 10, with higher scores indicating worse distress.
  Prior to administration of the distress thermometer measure, each caregiver will be asked if they are experiencing distress related to Covid-19 (yes/no). The distress thermometer asking them to rate their distress in the past week including today. The Covid-19 variable will be included as a covariate in the analyses.
  Evaluated for changes over 3 time points using repeated measures analysis of variance (RMANOVA)-between and within model- controlling for caregiver age, race, and gender

CONTACTS AND LOCATIONS:
Overall Officials: Sara Douglas, PhD, RN, Principal Investigator — Case Western Reserve University

IPD SHARING:
Plan to Share IPD: No
Pilot study